CLINICAL TRIAL: NCT01611246
Title: Performance of the Acclarent Iontophoresis System With Earset (IPSES) in Healthy Volunteers
Brief Title: Earset Healthy Volunteer Study
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Other Study IDs: CPR005031
Record Dates: First submitted 2012-05-29; First posted 2012-06-04 (Estimated); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anesthetization: Anesthetization
  Interventions: Device: Iontophoresis System With Earset

INTERVENTIONS:
Device: Iontophoresis System With Earset — iontophoresis of lidocaine-based solution for numbing tympanic membrane

SUMMARY:
The study will recruit healthy volunteers to undergo the Iontophoresis procedure using the Acclarent Iontophoresis System with Earset (IPSES).

ELIGIBILITY:
Inclusion Criteria:

* At least 12 months old

Exclusion Criteria:

* Pregnant or lactating females
* Subjects with history of sensitivity or reaction to lidocaine, tetracaine, epinephrine, or any hypersensitivity to local anesthetics of the amide type, or any component of the drug solution
* Significantly atrophic or perforated tympanic membrane
* Otitis externa
* Damaged or denuded skin in the auditory canal
* Electrically sensitive subjects and subjects with electrically sensitive support systems (pacemakers, defibrillators, etc.)
* Cerumen impaction resulting in a significant amount of cleaning required to visualize the tympanic membrane
* Evidence of Otitis Media at day of procedure, or within the past three (3) months prior to procedure.

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2012-08-01 (Actual); Study Completion 2012-08-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects anesthetized as assessed by Wong-Baker scale | Day 1

SECONDARY OUTCOMES:
Number of participants with serious adverse events | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Roberson, M.D., Principal Investigator — CEI Medical Group
Locations (1):
- CEI Medical Group, East Palo Alto, California, United States